CLINICAL TRIAL: NCT06859580
Title: Bisphosphonate vs. Placebo Prior to Parathyroidectomy in Primary Hyperparathyroidisme: A Randomized, Double-blinded Placebo-controlled Trial
Brief Title: Bisphosphonate Prior to Parathyroidectomy in Primary Hyperparathyroidism
Acronym: ZOLPHPT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZOLPHPT; 2024-520073-13-00 (EU CTIS Number); 2023-000007-39 (EudraCT Number)
Record Dates: First submitted 2025-02-25; First posted 2025-03-05 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: Primary Hyperparathyroidism
Keywords: zoledronate; parathyroidectomy; placebo
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — Zoledronic Acid; Saline Waters

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zoledronic acid (Active Comparator): Patients referred to Aarhus University Hospital (AUH) for PTX due to PHPT will be included prospectively. We aim to include 140 patients with PHPT - 70 patients in each group. Patients will be enrolled consecutively until the required number of participants have been achieved. Enrolled participants will be randomized to intervention (active medicine) or placebo group and receive either zoledronate or placebo (saline water) 2-4 weeks prior to PTX.
  Interventions: Drug: Zoledronic acid 4 mg
- Placebo (Placebo Comparator): Patients referred to Aarhus University Hospital (AUH) for PTX due to PHPT will be included prospectively. We aim to include 140 patients with PHPT - 70 patients in each group. Patients will be enrolled consecutively until the required number of participants have been achieved. Enrolled participants will be randomized to intervention (active medicine) or placebo group and receive either zoledronate or placebo (saline water) 2-4 weeks prior to PTX.
  Interventions: Drug: Natriumklorid 9 mg/ml, Fresenius Kabi

INTERVENTIONS:
Drug: Zoledronic acid 4 mg — Product name/EU MP number: Zoledronic Acid Oresund Pharma 4 mg/100 ml infusionsvätska, lösning/PRD8924813 (Test) Substance (name/ code): ZOLEDRONIC ACID/SUB00176MIG Strength: Zoledronic Acid 0.04mg Pharmaceutical form: SOLUTION FOR INFUSION Route of administration: INFUSIÓN INTRAVENOSA Marketing authorisation status (MA number, MS where authorised etc): 52486 / SE Modified in relation to MA: No Max Dosage: mg milligram(s) Duration of use: Week
  Other Names: ZOL; Zoledronate; Zoledronate acid
  Arms: Zoledronic acid
Drug: Natriumklorid 9 mg/ml, Fresenius Kabi — Product name/EU MP number: Natriumklorid "Baxter" ClearFlex 9 mg/ml,infusionsvæske, opløsning/PRD456031 (Placebo) Substance (name/ code): SODIUM CHLORIDE/SUB12581MIG Strength: Sodium Chloride 0.9g / 100mL Pharmaceutical form: SOLUTION FOR INFUSION Route of administration: INFUSIÓN INTRAVENOSA Marketing authorisation status (MA number, MS where authorised etc): 32466 / DK Modified in relation to MA: No Max Dosage: ml millilitre(s) Duration of use: Week
  Other Names: saline water
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blinded, placebo-controlled trial investigating the effects of zoledronic acid (ZOL) versus placebo in patients with primary hyperparathyroidism (PHPT) undergoing parathyroidectomy (PTX). PHPT is a common endocrine disorder associated with hypercalcemia, reduced bone mineral density (BMD), increased fracture risk, renal calcifications, and cardiovascular complications. While PTX remains the definitive treatment, the potential role of bisphosphonates in optimizing post-surgical outcomes remains unclear.

This trial aims to evaluate whether a single infusion of ZOL prior to PTX impacts bone health, cardiovascular parameters, and renal function one year post-surgery. The primary endpoint is the change in areal bone mineral density (aBMD) at the lumbar spine one year after PTX. Secondary endpoints include changes in aBMD at other skeletal sites, volumetric BMD, bone microarchitecture, bone turnover markers, coronary artery calcium score, arterial stiffness, and renal calcifications.

A total of 140 postmenopausal women and men over 50 years with PHPT and low BMD will be enrolled and randomized to receive either ZOL or placebo 2-4 weeks before PTX. Participants will undergo extensive imaging, biochemical analysis, and cardiovascular assessments at baseline and one year post-surgery.

This study seeks to clarify whether ZOL improves post-surgical bone recovery or interferes with the natural bone remodeling process following PTX. Additionally, it will provide insight into the cardiovascular and renal effects of bisphosphonate therapy in PHPT patients. Findings may help guide treatment strategies for optimizing long-term skeletal and systemic health in this patient population.

DETAILED DESCRIPTION:
Aim The overall aim of this study is a physiological investigation of the effect of bisphosphonate treatment versus placebo at time of parathyroidectomy (PTX) in patients with primary hyperparathyroidism (PHPT) on bone, kidney and the cardiovascular system one-year post-surgery.

Hypothesis:

In patients with PHPT and low areal bone mineral density (aBMD), treatment at time of PTX with zoledronic acid (ZOL) compared to placebo:

1. does not improve aBMD
2. does not improve bone microarchitecture
3. does not improve volumetric bone mineral density (vBMD)
4. does not influence changes in BTM
5. does not improve coronary artery calcium score (CACS)
6. does not improve arterial stiffness (pulse wave velocity [PWV])
7. does not improve degree of renal calcifications or urinary parameters

   Background:

   PHPT is a common endocrine disorder characterised by hypercalcemia and inappropriately high levels of parathyroid hormone (PTH). In most cases, PHPT is caused by hypersecretion of PTH from a single adenoma (80-90%). It is a chronic disease, which may lead to several complications such as osteoporosis, renal calcifications, cardiovascular disease, and neuropsychiatric symptoms. Surgical removal of the parathyroid gland/-s causing the hypersecretion of PTH is the only definitive cure for PHPT. It is a disease that mostly affects women with a ratio of 3:4 in the age group 40-70 years. Even though many patients are asymptomatic up to one third of the patients have osteoporosis at the time of diagnosis. Hypersecretion of PTH affects bone causing an increase in bone turnover markers (BTM), a decrease in BMD and an increased risk of fractures. Successful PTX normalises the calcium homeostasis and increases BMD one-year post-surgery at both lumbar spine and total hip, whereas the BMD increase at the distal forearm is minor. Accordingly, in Denmark, patients with PHPT and osteoporosis are most often treated with PTX only and "watchful waiting" is employed regarding BMD. If osteoporosis is sustained one year post surgery treatment (typically with a bisphosphonate) is, then initiated. To date, limited data on the effect of bisphosphonates if administrated at time of PTX is available. A retrospective study comparing 24 PHPT patients treated with PTX alone to 26 PHPT patients treated with both bisphosphonates and PTX found no beneficial effects on BMD of adding bisphosphonate to PTX. In another retrospective study however, co-treatment with bisphosphonate prior to PTX in patients with both PHPT and osteoporosis was associated with a decreased risk of fracture whereas, adding bisphosphonates after PTX did no reduce fracture risk. In contrast, a RCT in patients with PHPT comparing treatment with ZOL 1-3 months after PTX to PTX alone and found a significantly higher increase in BMD at the lumbar spine and femoral neck in the group treated with ZOL. At the total hip, however, BMD increased more in the group that only received PTX. Taken together the studies so far have shown conflicting results. Moreover, as the lumbar spine and femoral neck are sites relatively rich in trabecular bone with higher turn-over, whereas cortical bone is more prominent at the total hip, the effects of bisphosphonates and PTX may differ according to bone site. Therefore, it is unclear if treatment with bisphosphonate at time of PTX strengthens bone or impairs the natural recovery of bone during the first year after PTX. Only very few studies have addressed this issue. As up to one third of the patients with PHPT are diagnosed with osteoporosis, it is essential to clarify which treatment approach is optimal for the recovery of bone in this patient group. To clarify bisphosphonates effect on bone metabolism at the time of PTX, the investigators will perform a mechanistic study in patients with PHPT and either osteopenia or osteoporosis to study the pharmacodynamic effects on bone prior to PTX.

   Several studies have reported an increased mortality compared to the general population in patients with classic PHPT with moderate to severely elevated ionized calcium levels whilst studies with focus on mild PHPT found no increased mortality. Overall death was reported from cardiovascular diseases (CVD) and malignancy. ZOL is a well-known drug used for decades to treat osteoporosis and malignancy-related bone disease. However, possible positive effects such as reduced mortality and cardiovascular events of ZOL used have been discussed. In a RCT study investigating the effects of ZOL infusion every 18 months on BMD in postmenopausal women observed a lower rate of myocardial infarction and composite cardiovascular outcomes (defines as myocardial infarction, need for coronary revascularization, stroke or sudden dead) but not stroke in the group receiving ZOL compared to placebo. In contrast, meta-analyses looking at cardiovascular safety of ZOL , found no beneficial effects on major cardiovascular events with ZOL used, however, in one meta-analysis an increased risk of arterial fibrillation was observed.[22, 23] In a large cohort study from Denmark and Sweden investigating the safety of ZOL against oral bisphosphonate also observed a higher risk of atrial fibrillation, other arrhythmias, and heart failure compared to untreated individuals whereas the cardiovascular mortality among ZOL users was lower. Studies investigating effects of ZOL on cardiovascular outcomes are all made in population with osteoporosis or in patients with low BMD. However, no one have investigated ZOLs effect on cardiovascular indices in patients with PHPT. Coronary artery calcium score (CACS) and pulse wave velocity (PWV) are strong predictors of CVD in healthy individuals. Only few studies have investigated the CACS in PHPT patients. A cross-sectional study of 130 PHPT patients compared to a cohort of population-based control subjects found a greater positive CACS in PHPT patients compared to controls. However, another cross-sectional study of only 20 PHPT patients found no increased CACS compared to healthy controls.[28] Central arterial stiffness measured as PWV has been established as a predictor of cardiovascular events and all-cause mortality in both the middle-aged and elderly population. A few prospective studies have reported an increased arterial stiffness in PHPT patients compared to healthy individual and a decreased arterial stiffness following PTX. A RCT study investigating short-term effect of PTX on arterial stiffness observed a significant decrease in PWV 3-month after PTX in PHPT with moderate-severe hypercalcemia. As patients with PHPT have increased CVD mortality is it of great interest to investigated if ZOL infusion in PHPT may have a proactive effect on the cardiovascular system as well as beneficial effects on bone architecture.

   Renal calcifications are common in PHPT and in many studies the prevalence is determined to be around 20-25%. However, effects of PTX on the remission on renal calcifications are sparser. The risk of nephrolithiasis declines following PTX, although the risk remains increased compared to the general population. Hypercalciuria is of importance for the development of calcifications, however it does not fully explain the increased stone risk. Other metabolic factors in the urine may play a role in the increased risk of renal calcifications. One study with 51 PHPT patients found normalization of urinary calcium excretion following PTX but not on all other urinary metabolic parameters. As only few studies have evaluated the effect of PTX on urinary parameters and renal calcifications one-year post-surgery the investigators want to assess a metabolic urinary profile and a CT-scan of the kidneys and urinary tracts in PHPT with renal calcifications compared to PHPT without calcifications and effects of PTX as well as the potential effects of treatment with ZOL.

   Methods Design: A randomized, double-blinded placebo-controlled trial

   Patient flow: Patients referred to Aarhus University Hospital (AUH) for PTX due to PHPT will be included prospectively. The investigators aim to include 140 patients with PHPT - 70 patients in each group. Patients will be enrolled consecutively until the required number of participants have been achieved. The enrolment period will be approximately 1 years. Enrolled participants will be randomized to intervention- or placebo group and receive either ZOL or placebo (saline water) 2-4 weeks prior to PTX. Enrolled participants will be examined as detailed below (table 1). Participants who did not archive normocalcemia following PTX may not have to continue their participation in the study after (unsuccessful) PTX. One-year post-surgery a control visit will be held for all participants. The participants finish the study at the 12- month follow-up visit after PTX. Participants will be excluded from the study if a ionized calcium >1,35 mmol/l is measured at day 28.

   Intervention:

   ZOL 4 mg vs. placebo (100 ml saline water) as a single intravenous (iv) infusion. Participants will receive ZOL or saline water at the outpatient clinic of Endocrinology, Aarhus University Hospital approximately two-four weeks prior to PTX (baseline). According to standard of care at the hospital, all patients will be recommended a daily oral supplement with 800 mg of elementary calcium in combination with 38 micrograms of cholecalciferol following PTX.

   Double blinding: A nurse with no association to the project will mask both ZOL and saline water prior to randomisation with non-transparent bags so that both patients and investigators in the trial are blinded to the content of the infusion bags. At time of inclusion, participants will be randomised (double blinded) to receive either ZOL or placebo (saline) 2-4 weeks prior to PTX. ZOL and saline water will be administrated as an iv. infusion over 15 minutes by a study nurse without any other relation to the study. Randomization will be performed using a computer algorithm. Overall, participants will be stratified based on gender and ionized calcium ≤ or ≥ 1,45 mmol/l into 2 approximately equally sized groups. One of the groups will also have BTM performed at day 14 and at week 8, 16 and 24.

   Overall medical records:

   ZOL and placebo (saline water) are supplied by the hospital pharmacy and delivered to the investigation site. The investigators will document and keep a record of experimental drug delivered to the site with the following information: name, strength, amount received, date of receipt, batch number, expiration date, amount of experimental drug on the investigation site, date and initials on the person which has updated the records of the experimental drug delivered. The delivery note from the pharmacy may be used as documentations provided it contains the above information and will be signed upon receipt.

   Individual medical records:

   Medical records for each participant will be carried out thoroughly. A separate document will be used for the individual medical records to obtain blinding. Before the experimental drug is delivered to the investigator a second person with no association to the project will double check that is it the correct experimental drug delivered to the investigator according to the randomisation. The medical records will contain the following information: Patients ID, name, strength, and amount of the experimental drug, batch number, expiration date, amount of drug delivered and administered, date and initials of persons delivered and administrated the drug, amount of experimental drug returned, date and initial of person receiving returned experimental drug.

   Unblinding:

   The investigator has the responsibility and the possibility to unblind participants in case of emergency.

   Measurements:

   aBMD are measured by dual energy x-ray absorptiometry (DXA) and high-resolution peripheral computed tomography (HRpQCT) scans at baseline and end of study. Volumetric bone mineral density is measured by bone assessment included in the Cardiac CT-scan (see below). Biochemistry includes blood teste of plasma levels of PTH, vitamin D metabolites (including 25-hydroxyvitamin D [25(OH)D] and calcitriol [1,25(OH)2D]), total and ionized calcium (Ca2+), phosphate, magnesium, albumin, sodium, potassium, creatinine, estimated glomerular filtration rate (eGFR), cystatin C (CysC), aldosterone, renin, angiotensin 2, arginine vasopressine, insulin, glucose, glycated HbA1c, total cholesterol, low density lipoprotein (LDL), high-density lipoprotein (HDL) and triglycerides.

   At some time points blood is also analyzed in terms of a "BTM package" which includes analyses for C-terminal telopeptide of type I collagen [CTX], N-terminal propeptide of type I procollagen [PINP], bone specific alkaline phosphatase [BSAP]), and fibroblast growth factor 23 [FGF-23] as well as analyses of plasma Ca2+ and creatinine. In approximately half of the participants (who accept extended BTM measurements), BTM are also measured after 2 weeks and after approximately 2, 4 and 6 months (Table 1).

   In 24-hour urine, volume is measured, and the urine is analyzed for excretion of calcium, phosphate, sodium, potassium, magnesium, oxalate, uric acid and citrate.

   Some analyses are performed in batches for which samples will be frozen in a research biobank and not analyzed before all samples have been collected which includes PTH, vitamin D metabolites, BTM, insulin, aldosterone, renin, angiotensin 2, arginine vasopressine and CysC as well as urinary citrate.

   Cardiac CT-scan is performed at the Department of Cardiology at Gødstrup Regional Hospital and will include the heart, kidney and proximal femur. A cardiac ultrasound (ECHO) will be performed together with the CT-scan. An eGFR ≥ 35 mL/min must be measured within three months prior to the scan. Otherwise, a blood sample will be performed prior to the scan or on the day. From the Cardiac CT-scan the coronary artery plaque burden will be measured as a CAC-score. Furthermore, the CT-scan will provide data on vBMD at the lumbar spine and hip, vertebral compression fractures and renal calcifications.

   Tonometry: The SphygmoCor system (Xcel; AtCor Medical, Sydney, NSW, Australia) is an ultrasound examination used to assess arterial stiffness and pulse wave analysis (PWA). For measurements of PWV an inflated femoral cuff will be placed on the right-upper thigh combined with carotid applanation tonometry.

   Questionnaires: Parathyroid assessment of symptoms score (PAS) and primary hyperparathyroidism health related quality of life (PHPQoL) will be handed out at baseline and at 12-month follow-up. Furthermore, all participants will receive a questionnaire about possible side-effects to infusion 1-week and one month after receiving either ZOL or placebo (attachment 1).

   Statistics: Assuming a mean BMD of 0.9 g/cm2 at the lumbar spine and an estimated differences of 2% in BMD between groups one year after surgery (5% significant level, 90% power, SDdiff 0.03 g/cm2) 59 participants are needed in each group. To accounts for dropouts 70 participants will be included in each group. QQ-plots will be used to check for normality. The difference between the two groups will be assessed using either a paired t-test or Mann-Whitney U-test depending on distribution for continuous variables. The investigators will use intention to treat analysis including all randomized participants with a successful PTX (i.e., analysis will be restricted to participants archiving normocalcemia following surgery).

   Side effects
   1. Intervention ZOL is a well-known drug that has been used for many years in treating osteoporosis and other metabolic bone diseases. It is well tolerated. However, there are some known side effects. Some participants may experience fever and muscle pain after infusion of ZOL (flu like symptoms). The side effects are benign, last only a few days and discomfort can be reduced by administration of paracetamol. Furthermore, some participants may experience joint pain which often disappear again after weeks. Allergy towards bisphosphonate is a very rare and an uncommon side effect. ZOL acid given as a single infusion is not expected to give any long-term side effects. Furthermore, infusion of 100 ml of saline water is not expected to give any short- or long-term side effects.
   2. Other side effects During the project, less than 300 mL of full blood will be drawn and should not give any unpleasantness for the participants. Furthermore, to infuse ZOL or saline water an i.v. access is necessary. However, some may find it uncomfortable to have a blood test taken and an i.v. access established. There is only a minimal risk of infection at the injection sites.

   The cardiac CT is implemented in everyday clinical work, and to evaluate possible coronary stenosis it includes a contrast-enhanced sequence with an iodine agent. Participants' renal function is evaluated with a blood sample prior to the scan (e-GFR ≥ 35 ml/min/1.73 m3) for safety reasons. Furthermore, in very rare cases, participants develop an allergic reaction to iodine contrast and therefore participants are asked about prior allergic reactions to iodine before the CT scan. Moreover, a medical doctor will be present during the CT scan.

   Betablockers (atenolol administered orally 30 min-2 hours before the scan or metoprolol administered intravenously during the scan) or ivabradine (administered orally 30 min-2 hours before the scan) are used to lower the heart rate during the cardiac CT. Likewise, a vasodilator (nitroglycerin) is administered sublingually immediately prior to the scan. Both betablockers, ivabradine, and nitro-glycerine are administered to lower radiation doses and improve image quality. This standard procedure is also used in a clinical setting, and it is considered safe. The potential side effects are nausea, headache, dizziness, abdominal pain, or obstipation, and are considered minimal and short term. A medical doctor with experience in cardiac CT will evaluate the scans for critical cardiac disease (defined as a >50% stenosis in left main coronary artery (CT angiography) or left ventricular ejection fraction below 30% by ECHO).

   Each CT-scan will cause a radiation of 10.0 mSv which corresponds to 3 years of background radiation. DXA- and HRpQCT scans are without discomfort for the patients. At each DXA-scan patient receive a total radiation dose of maximal 0.2 mSV which correspond to 30 days of background radiation. At each HRpQCT scan, a patient receives a total radiation dose of maximal 0.003 mSV which correspond to less than one day of background radiation.

   Accordingly, at baseline each patient will receive a total dose slightly higher than 10.2 mSv corresponding to 3.1 years of background radiation. As the examinations are repeated after one year, the total radiation will correspond to 6,2 years of background radiation and increase the risk of dying from cancer from 25.0% to 25.1%. However, the actual risk is probably less, as this study is performed in an elderly population (all > 50 years of age) with an estimated median age of 64 years. As the investigation will provide important information on whether surgery should be encouraged in this patient population and the presence of potential debilitating comorbidities that require attention and further treatment, this risk is considered as reasonable, and the investigators believe the potential gains from this study outweigh the risks.

   Tonometry and ECHO are non-invasive procedures using ultrasound, and no direct harm or discomfort is caused to the participants.

   Management of incidents and side effects Product summary for ZOL will be used as a reference document in case of side effects. All adverse events (suspected or unsuspected) will be documented in case report forms (CRF) and handled in accordance with the general practice of the hospital. Registration of incident and side effects starts at the initiation of experimental drug for each participant and ends at the last control visit 12-month post-surgery. The participants will therefore be followed for approximately 12-13 months after administration of the experimental drug (which is administrated 2-4 weeks before surgery).

   Definition in according to the notice for clinical trials are:
   * Incident: Any adverse incident in a patient or a participant in a clinical trial after treatment with a medical product without there necessarily being a connection between this treatment and the adverse incident.
   * Side effect: Any harmful and unwanted reaction to an investigational drug regardless of the dose. A side effect that is inconsistent with the product information.
   * Seriously incident and side effects: An incident or side effect that regardless of the dose results in death, is life-threatening, entails hospitalization or prolongation of hospital stay, which results in significant or permanent disability or leads to a congenital anomaly or deformity.

   It is the investigator who has the responsibility to investigate and evaluate reported incidences and assess whether these incidences are adverse reactions (AR) or adverse events (SAR). Within 24 hours the investigator must report all serious incidences/side effects to sponsor.

   Sponsor will immediately report to EudraVigilance in case of any suspected unexpected serious adverse reactions (SUSAR). Sponsor must ensure that all SUSAR that are life threatening or deadly/results in dead are registered and reported to EudraVigilance as soon as possible and no later than 7 days after the SUSAR is registered. All other SUSAR must be reported to EudraVigilance no later than 15 days after the SUSAR has been registered. It is the sponsor who evaluate whether a seriously incidence/side effect is expected, or none expected according to the product resume and thereby a SUSAR or an expected seriously incidence/side effect. SUSARs will be reported electronically to the SUSAR database (EudraVigilance Clinical Trial Module E2B) using the e-form.

   Once a year throughout the trial period, the sponsor must prepare a list of all serious suspected adverse events (SAR) that occurred during the trial period and a report on the safety of the participants. The list and reports will be submitted to the competent authorities, i.e., the EU Clinical Trial Information System (CTIS) and The Central Denmark Region Committees on Health Research Ethics.

   End of trial:

   Results of the trial will be reported in EudraCT as soon as possible and no later than one year after the end of the trial.

   Research biobank Only blood and urine are collected. Approximately 300 ml of full blood will be drawn from the participants during the 1 year of trial which will be used for biochemical analyses. Collected biological material will be stored in a research biobank, under the premise of written consent from the participant. Blood samples are collected using standard methods and stored in a freezer (-20/-80C). Analysis will be carried out at the end of the study at the Department of Biochemistry, Aarhus University Hospital. At the end of the project excessive biological material will be transferred to a biobank for future research. It will generally require a new consent if excessive biological material is used for other research in the future. Furthermore, new research on excessive biological material will be reported to the Central Denmark Region Committees on Health Research Ethics.

   Clinical data The following information will be disclosed from the medical chart to the research project: Patient demography, co-morbidities, use of medications, smoking history and use of alcohol, indication for surgery, fracture history, results of DXA scan, X-ray of the spine, and CT scans of the kidneys and urinary tracts, histological diagnosis of the resected parathyroid gland/-s and the following biochemistry; P-PTH, P-ionized and total calcium, P-phosphate, P-magnesium, P-alkaline phosphatase, P-albumin, P-creatinine, estimated glomerular filtration rate (eGFR), 1,25-dihydroxyvitamin-D and 25-hydroxyvitamin-D. This information will be used to validate the diagnosis and possible complications following PHPT.

   Economics The trial is initiated by the applicants. Financial support has been granted by the Novo Nordic Foundation and additional support will be applied for from public and private funds. Financial support will be used to cover medical expensive and remuneration of staff.

   Recruitment Patients fulfilling the inclusion criteria will be enrolled after oral and written informed consent. Patients will be thoroughly informed about effects and possible side effects of ZOL. Patients will be approached by medical doctors either at the Department of Endocrinology and Internal Medicine, AUH during their diagnostic work-up for PHPT or during their appointment about PTX at the Department of Oto-Rhino-Laryngology, AUH. The conversation will be held behind closed doors. If a participant wants an assistant during the interview the meeting can be rescheduled on a following day. Possible participants have up to 2 weeks to decide.

   Publications The investigators will aim to publish results from this project - negative, positive, as well as inconclusive results in international peer reviewed journals.

   Ethical aspects Participants will be informed thoroughly about the project's aim, execution, and possible side effects both orally and in written. The project is voluntarily, and the participants can withdraw their consent anytime during the project. If a participants decide to withdraw, it will not affect their ongoing and future treatments. Participants will only be enrolled in the project by given full consent orally and in written. ZOL is a well-known drug that have been used for many years in treatment of osteoporosis. Typical side-effects observed after a single dose are often mild and transitory. Long-term side effects are not expected after a single dose of ZOL. Placebo (100 ml of saline water) is used in the project of methodological reasons. All patients enrolled in the project will all undergo PTX and therefore receive treatment for their hyperparathyroid hypercalcemia without any delays.

   If the investigators find signs of unknown diseases including critical coronary artery disease or severe heart failure, participants will be offered further investigation and/or treatment. Image-based findings unrelated to the heart, kidneys (excluding adrenal glands), and spine will not be a part of the study, and this will be stated in the participant information. In prior studies, single participants were diagnosed with lung cancer after their participation in the screening and a retrospective evaluation of CT images revealed that the cancer disease could have been observed at an earlier stage. This has led to a principal evaluation at the Danish Agency for Patient Complaints (file number: 2018-3464) and the Board of Appeal (file number 2019-6646), which both concluded that no criticism could be held against the study.

   CAC measurements may be useful to optimizing CVD risk stratification by identifying persons with undiagnosed subclinical disease, who should receive multifactorial intensified preventive treatment, but also to identify true low-risk persons in whom reduction of expensive medication with potential side-effects would be appropriate.

   Clauses There are no clauses to inform.

   Insurance The project is covered by Aarhus University Hospital patient insurance.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal females or males > 50 years
2. A diagnosis of hyperparathyroid hypercalcemia due to sporadic PHPT referred to PTX
3. aBMD T-score ≤ -1 at total hip, femoral neck, or lumbar spine
4. 25-hydroxyvitamin D ≥ 50 nmol/l prior to randomization
5. Willingness to undergo PTX

Exclusion Criteria:

1. Known or suspected familial ethology (e.g., MEN1 or 2)
2. Estimated glomerular filtration rate < 35 ml/min
3. Known allergy to bisphosphonates
4. Planned or recent (within the last 3 months) major dental procedures (e.g., jaw surgery or tooth extraction)
5. Chronic or acute disorders (e.g., rheumatoid arthritis, inflammatory bowel disease, cancer) or prior medications (e.g., lithium, glucocorticoids within the last year, antiresorptive or bone anabolic treatment within the last 3 years) known to affect bone metabolism.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Effects of ZOL vs. placebo at time of parathyroidectomy based on change in aBMD at lumbar spine meased at baseline compared to one year after PTX. | 12 months (one year)
  aBMD (g/cm^3) will be measured by DXA-scans at baseline and one year after PTX.

SECONDARY OUTCOMES:
Effects of ZOL at aBMD at distal forearm | 12 months (one year)
  A change in aBMD (g/cm^3) at distal forearm will be measured by DXA-scans at baseline and 12 month after PTX.
Effects of ZOL at aBMD at femoral neck | 12 months (one year)
  A change in aBMD (g/cm^3) at femoral neck will be measured by DXA-scans at baseline and 12 month after PTX.
Effects of ZOL at aBMD at total hip | 12 months (one year)
  A change in aBMD (g/cm^3) at total hip will be measured by DXA-scans at baseline and 12 month after PTX.
Effects on microarchitecture measured by high-resolution peripheral computed tomography (HRpQCT). | 12 months
  Bone microarchitecture will be measured by HRPqCT scans and changes will be assessed from baseline to 12 months after PTX.
Effects on biochemical bone turnover markers (BTM). | 12 months
  Blood samples will be drawn from participants and analyses of bone turnover markers (CTx, P1NP, BSAP and FGF-23) at baseline, 7 and 28 days after parathyroidectomy and 12 months after PTX will be performed.
Effects on vBMD at the hip | 12 months
  The investigators will perform CT-scans of the hip at baseline and after 12 months in those patients who are accepting extra CT-scans.
Effects on vBMD at the lumbar spine. | 12 months
  The investigators will perform CT-scans of the lumbar spine at baseline and after 12 months in those patients who are accepting extra CT-scans.
Effects on coronary artery calcium score (CACS) | 12 months
  Heart CT-scans will be performed in those patients who accept this at baseline and 12 months after PTX and analyse CACS (from 0 to 10.000) in these patients.
Effects on pulse wave velocity (PWV) | 12 months
  Tonometry will be performed and a measure of PWV (measured as m/s) will be analysed at baseline and 12 months after PTX.
Effects of ZOL on renal calcifications | 12 months
  The investigators will perform CT-scans of the kidneys for those participants who accepts this scan at baseline and 12 months after PTX.
Effects of ZOL on urinary analytes | 12 months
  The investigators will examine 24-hour urine, which will be analyzed for excretion of calcium, phosphate, sodium, potassium, magnesium, oxalate, uric acid and citrate at baseline and 12 months after PTX.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Rejnmark, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus N, Central Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, CSR
Time Frame: Start date is time of publication. End date is 5 years after publication.
Access Criteria: By contacting the leading author of the publication in order to make a data sharing agreement, which should be signed. Proposal for agreement must contain planned analyses. Statistical analyses have to be approved by independent review before published. Data sharing agreement needs to be approved by the Technology Transfer Office (TTO), Aarhus University Hospital, Denmark.

REFERENCES:
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Marchini GS, Faria KVM, Torricelli FCM, Monga M, Srougi M, Nahas WC, Mazzucchi E. Sporadic primary hyperparathyroidism and stone disease: a comprehensive metabolic evaluation before and after parathyroidectomy. BJU Int. 2018 Feb;121(2):281-288. doi: 10.1111/bju.14072. Epub 2017 Nov 28. PMID 29124877
- [Background] Odvina CV, Sakhaee K, Heller HJ, Peterson RD, Poindexter JR, Padalino PK, Pak CY. Biochemical characterization of primary hyperparathyroidism with and without kidney stones. Urol Res. 2007 Jun;35(3):123-8. doi: 10.1007/s00240-007-0096-2. Epub 2007 May 3. PMID 17476495
- [Background] Frokjaer VG, Mollerup CL. Primary hyperparathyroidism: renal calcium excretion in patients with and without renal stone sisease before and after parathyroidectomy. World J Surg. 2002 May;26(5):532-5. doi: 10.1007/s00268-001-0262-6. Epub 2002 Feb 19. PMID 12098039
- [Background] Corbetta S, Baccarelli A, Aroldi A, Vicentini L, Fogazzi GB, Eller-Vainicher C, Ponticelli C, Beck-Peccoz P, Spada A. Risk factors associated to kidney stones in primary hyperparathyroidism. J Endocrinol Invest. 2005 Feb;28(2):122-8. doi: 10.1007/BF03345354. PMID 15887857
- [Background] Deaconson TF, Wilson SD, Lemann J Jr. The effect of parathyroidectomy on the recurrence of nephrolithiasis. Surgery. 1987 Dec;102(6):910-3. PMID 3686354
- [Background] Mollerup CL, Vestergaard P, Frokjaer VG, Mosekilde L, Christiansen P, Blichert-Toft M. Risk of renal stone events in primary hyperparathyroidism before and after parathyroid surgery: controlled retrospective follow up study. BMJ. 2002 Oct 12;325(7368):807. doi: 10.1136/bmj.325.7368.807. PMID 12376441
- [Background] Mollerup CL, Lindewald H. Renal stones and primary hyperparathyroidism: natural history of renal stone disease after successful parathyroidectomy. World J Surg. 1999 Feb;23(2):173-5; discussion 176. doi: 10.1007/pl00013175. PMID 9880427
- [Background] Cooperberg MR, Duh QY, Stackhouse GB, Stoller ML. Oral calcium supplementation associated with decreased likelihood of nephrolithiasis prior to surgery for hyperparathyroidism. Int J Urol. 2007 Dec;14(12):1113-5. doi: 10.1111/j.1442-2042.2007.01904.x. PMID 18036056
- [Background] Moosgaard B, Vestergaard P, Heickendorff L, Melsen F, Christiansen P, Mosekilde L. Vitamin D status, seasonal variations, parathyroid adenoma weight and bone mineral density in primary hyperparathyroidism. Clin Endocrinol (Oxf). 2005 Nov;63(5):506-13. doi: 10.1111/j.1365-2265.2005.02371.x. PMID 16268801
- [Background] Starup-Linde J, Waldhauer E, Rolighed L, Mosekilde L, Vestergaard P. Renal stones and calcifications in patients with primary hyperparathyroidism: associations with biochemical variables. Eur J Endocrinol. 2012 Jun;166(6):1093-100. doi: 10.1530/EJE-12-0032. Epub 2012 Apr 3. PMID 22474170
- [Background] Ejlsmark-Svensson H, Bislev LS, Rolighed L, Sikjaer T, Rejnmark L. Predictors of Renal Function and Calcifications in Primary Hyperparathyroidism: A Nested Case-Control Study. J Clin Endocrinol Metab. 2018 Sep 1;103(9):3574-3583. doi: 10.1210/jc.2018-00923. PMID 29955845
- [Background] Ejlsmark-Svensson H, Rolighed L, Rejnmark L. Effect of Parathyroidectomy on Cardiovascular Risk Factors in Primary Hyperparathyroidism: A Randomized Clinical Trial. J Clin Endocrinol Metab. 2019 Aug 1;104(8):3223-3232. doi: 10.1210/jc.2018-02456. PMID 30860588
- [Background] Rosa J, Raska I Jr, Wichterle D, Petrak O, Strauch B, Somloova Z, Zelinka T, Holaj R, Widimsky J Jr. Pulse wave velocity in primary hyperparathyroidism and effect of surgical therapy. Hypertens Res. 2011 Mar;34(3):296-300. doi: 10.1038/hr.2010.232. Epub 2010 Nov 25. PMID 21107330
- [Background] Schillaci G, Pucci G, Pirro M, Monacelli M, Scarponi AM, Manfredelli MR, Rondelli F, Avenia N, Mannarino E. Large-artery stiffness: a reversible marker of cardiovascular risk in primary hyperparathyroidism. Atherosclerosis. 2011 Sep;218(1):96-101. doi: 10.1016/j.atherosclerosis.2011.05.010. Epub 2011 May 18. PMID 21645899
- [Background] Cansu GB, Yilmaz N, Ozdem S, Balci MK, Suleymanlar G, Arici C, Boz A, Sari R, Altunbas HA. Parathyroidectomy in asymptomatic primary hyperparathyroidism reduces carotid intima-media thickness and arterial stiffness. Clin Endocrinol (Oxf). 2016 Jan;84(1):39-47. doi: 10.1111/cen.12952. Epub 2015 Oct 12. PMID 26399562
- [Background] Streeten EA, Munir K, Hines S, Mohamed A, Mangano C, Ryan KA, Post W. Coronary artery calcification in patients with primary hyperparathyroidism in comparison with control subjects from the multi-ethnic study of atherosclerosis. Endocr Pract. 2008 Mar;14(2):155-61. doi: 10.4158/EP.14.2.155. PMID 18308652
- [Background] Koubaity O, Mandry D, Nguyen-Thi PL, Bihain F, Nomine-Criqui C, Demarquet L, Croise-Laurent V, Brunaud L. Coronary artery disease is more severe in patients with primary hyperparathyroidism. Surgery. 2020 Jan;167(1):149-154. doi: 10.1016/j.surg.2019.05.094. Epub 2019 Oct 24. PMID 31668778
- [Background] Townsend RR. Arterial stiffness and chronic kidney disease: lessons from the Chronic Renal Insufficiency Cohort study. Curr Opin Nephrol Hypertens. 2015 Jan;24(1):47-53. doi: 10.1097/MNH.0000000000000086. PMID 25470015
- [Background] Meyer M, Henzler T, Fink C, Vliegenthart R, Barraza JM Jr, Nance JW Jr, Apfaltrer P, Schoenberg SO, Wasser K. Impact of coronary calcium score on the prevalence of coronary artery stenosis on dual source CT coronary angiography in caucasian patients with an intermediate risk. Acad Radiol. 2012 Nov;19(11):1316-23. doi: 10.1016/j.acra.2012.06.006. Epub 2012 Aug 14. PMID 22897947
- [Background] Rubin KH, Moller S, Choudhury A, Zorina O, Kalsekar S, Eriksen EF, Andersen M, Abrahamsen B. Cardiovascular and skeletal safety of zoledronic acid in osteoporosis observational, matched cohort study using Danish and Swedish health registries. Bone. 2020 May;134:115296. doi: 10.1016/j.bone.2020.115296. Epub 2020 Feb 22. PMID 32097760
- [Background] Liu S, Tan Y, Huang W, Luo H, Pan B, Wu S. Cardiovascular safety of zoledronic acid in the treatment of primary osteoporosis: A meta-analysis and systematic review. Semin Arthritis Rheum. 2024 Feb;64:152304. doi: 10.1016/j.semarthrit.2023.152304. Epub 2023 Nov 8. PMID 37984227
- [Background] Kranenburg G, Bartstra JW, Weijmans M, de Jong PA, Mali WP, Verhaar HJ, Visseren FLJ, Spiering W. Bisphosphonates for cardiovascular risk reduction: A systematic review and meta-analysis. Atherosclerosis. 2016 Sep;252:106-115. doi: 10.1016/j.atherosclerosis.2016.06.039. Epub 2016 Jun 24. PMID 27513349
- [Background] Reid IR, Horne AM, Mihov B, Stewart A, Garratt E, Bastin S, Gamble GD. Effects of Zoledronate on Cancer, Cardiac Events, and Mortality in Osteopenic Older Women. J Bone Miner Res. 2020 Jan;35(1):20-27. doi: 10.1002/jbmr.3860. Epub 2019 Oct 11. PMID 31603996
- [Background] Billington EO, Reid IR. Benefits of Bisphosphonate Therapy: Beyond the Skeleton. Curr Osteoporos Rep. 2020 Oct;18(5):587-596. doi: 10.1007/s11914-020-00612-4. PMID 32734512
- [Background] Palmer M, Adami HO, Bergstrom R, Jakobsson S, Akerstrom G, Ljunghall S. Survival and renal function in untreated hypercalcaemia. Population-based cohort study with 14 years of follow-up. Lancet. 1987 Jan 10;1(8524):59-62. doi: 10.1016/s0140-6736(87)91906-4. PMID 2879173
- [Background] Ogard CG, Engholm G, Almdal TP, Vestergaard H. Increased mortality in patients hospitalized with primary hyperparathyroidism during the period 1977-1993 in Denmark. World J Surg. 2004 Jan;28(1):108-11. doi: 10.1007/s00268-003-7046-0. Epub 2003 Dec 4. PMID 14648050
- [Background] Hedback G, Tisell LE, Bengtsson BA, Hedman I, Oden A. Premature death in patients operated on for primary hyperparathyroidism. World J Surg. 1990 Nov-Dec;14(6):829-35; discussion 836. doi: 10.1007/BF01670531. PMID 2256355
- [Background] Ryhanen EM, Koski AM, Loyttyniemi E, Valimaki MJ, Kiviniemi U, Schalin-Jantti C. Postoperative zoledronic acid for osteoporosis in primary hyperparathyroidism: a randomized placebo-controlled study. Eur J Endocrinol. 2021 Aug 27;185(4):515-524. doi: 10.1530/EJE-21-0322. PMID 34324430
- [Background] Orr LE, Zhou H, Zhu CY, Haigh PI, Adams AL, Yeh MW. Skeletal effects of combined medical and surgical management of primary hyperparathyroidism. Surgery. 2020 Jan;167(1):144-148. doi: 10.1016/j.surg.2019.04.059. Epub 2019 Sep 30. PMID 31582307
- [Background] Lee IT, Sheu WH, Tu ST, Kuo SW, Pei D. Bisphosphonate pretreatment attenuates hungry bone syndrome postoperatively in subjects with primary hyperparathyroidism. J Bone Miner Metab. 2006;24(3):255-8. doi: 10.1007/s00774-005-0680-x. PMID 16622740
- [Background] Choe HJ, Koo BK, Yi KH, Kong SH, Kim JH, Shin CS, Chai JW, Kim SW. Skeletal effects of combined bisphosphonates treatment and parathyroidectomy in osteoporotic patients with primary hyperparathyroidism. J Bone Miner Metab. 2022 Mar;40(2):292-300. doi: 10.1007/s00774-021-01279-2. Epub 2021 Nov 10. PMID 34761302
- [Background] Sankaran S, Gamble G, Bolland M, Reid IR, Grey A. Skeletal effects of interventions in mild primary hyperparathyroidism: a meta-analysis. J Clin Endocrinol Metab. 2010 Apr;95(4):1653-62. doi: 10.1210/jc.2009-2384. Epub 2010 Feb 3. PMID 20130069
- [Background] Vestergaard P, Mollerup CL, Frokjaer VG, Christiansen PM, Blichert-Toft M, Mosekilde L. [Cohort study of fracture risk before and after surgery of primary hyperparathyroidism]. Ugeskr Laeger. 2001 Sep 3;163(36):4875-8. Danish. PMID 11571864
- [Background] Rolighed L, Vestergaard P, Heickendorff L, Sikjaer T, Rejnmark L, Mosekilde L, Christiansen P. BMD improvements after operation for primary hyperparathyroidism. Langenbecks Arch Surg. 2013 Jan;398(1):113-20. doi: 10.1007/s00423-012-1026-5. Epub 2012 Nov 7. PMID 23132462
- [Background] Melton LJ 3rd, Atkinson EJ, O'Fallon WM, Heath H 3rd. Risk of age-related fractures in patients with primary hyperparathyroidism. Arch Intern Med. 1992 Nov;152(11):2269-73. PMID 1444687
- [Background] Lundstam K, Heck A, Godang K, Mollerup C, Baranowski M, Pernow Y, Aas T, Hessman O, Rosen T, Nordenstrom J, Jansson S, Hellstrom M, Bollerslev J; SIPH Study Group. Effect of Surgery Versus Observation: Skeletal 5-Year Outcomes in a Randomized Trial of Patients With Primary HPT (the SIPH Study). J Bone Miner Res. 2017 Sep;32(9):1907-1914. doi: 10.1002/jbmr.3177. Epub 2017 Jul 7. PMID 28543873
- [Background] Khosla S, Melton LJ 3rd, Wermers RA, Crowson CS, O'Fallon Wm, Riggs Bl. Primary hyperparathyroidism and the risk of fracture: a population-based study. J Bone Miner Res. 1999 Oct;14(10):1700-7. doi: 10.1359/jbmr.1999.14.10.1700. PMID 10491217
- [Background] Kenny AM, MacGillivray DC, Pilbeam CC, Crombie HD, Raisz LG. Fracture incidence in postmenopausal women with primary hyperparathyroidism. Surgery. 1995 Jul;118(1):109-14. doi: 10.1016/s0039-6060(05)80017-0. PMID 7604371
- [Background] Ejlsmark-Svensson H, Rolighed L, Harslof T, Rejnmark L. Risk of fractures in primary hyperparathyroidism: a systematic review and meta-analysis. Osteoporos Int. 2021 Jun;32(6):1053-1060. doi: 10.1007/s00198-021-05822-9. Epub 2021 Feb 1. PMID 33527175
- [Background] Christiansen P, Steiniche T, Brixen K, Hessov I, Melsen F, Heickendorff L, Mosekilde L. Primary hyperparathyroidism: effect of parathyroidectomy on regional bone mineral density in Danish patients: a three-year follow-up study. Bone. 1999 Nov;25(5):589-95. doi: 10.1016/s8756-3282(99)00207-0. PMID 10574580
- [Background] Christiansen P, Steiniche T, Brixen K, Hessov I, Melsen F, Charles P, Mosekilde L. Primary hyperparathyroidism: biochemical markers and bone mineral density at multiple skeletal sites in Danish patients. Bone. 1997 Jul;21(1):93-9. doi: 10.1016/s8756-3282(97)00078-1. PMID 9213014
- [Background] Fraser WD. Hyperparathyroidism. Lancet. 2009 Jul 11;374(9684):145-58. doi: 10.1016/S0140-6736(09)60507-9. PMID 19595349
- [Background] Ejlsmark-Svensson H, Bislev LS, Lajlev S, Harslof T, Rolighed L, Sikjaer T, Rejnmark L. Prevalence and Risk of Vertebral Fractures in Primary Hyperparathyroidism: A Nested Case-Control Study. J Bone Miner Res. 2018 Sep;33(9):1657-1664. doi: 10.1002/jbmr.3461. Epub 2018 Jun 7. PMID 29734476